CLINICAL TRIAL: NCT03367793
Title: Identification of Optimum Spectacle Prescriptions for Patients With Down Syndrome
Brief Title: Spectacles for Patients With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Heather A. Anderson, Associate Professor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EY024590
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Vision, Low
MeSH Terms: conditions — Vision, Low | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Clinical, then Metric #1, then Metric #2 (Experimental): Each subject will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the clinically derived prescription first, followed by the metric-derived #1, and lastly the metric-derived #2.
  Interventions: Device: Spectacles - Clinically Derived; Device: Spectacles - Metric Technique #1 Derived; Device: Spectacles - Metric Technique #2 Derived
- Clinical, then Metric #2, then Metric #1 (Experimental): Each subject will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the clinically derived prescription first, followed by the metric-derived #2, and lastly the metric-derived #1.
  Interventions: Device: Spectacles - Clinically Derived; Device: Spectacles - Metric Technique #1 Derived; Device: Spectacles - Metric Technique #2 Derived
- Metric #1, then Clinical, then Metric #2 (Experimental): Each subject will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #1 prescription first, followed by the clinically derived prescription, and lastly the metric-derived #2 prescription.
  Interventions: Device: Spectacles - Clinically Derived; Device: Spectacles - Metric Technique #1 Derived; Device: Spectacles - Metric Technique #2 Derived
- Metric #2, then Clinical, then Metric #1 (Experimental): Each subject will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #2 prescription first, followed by the clinically derived prescription, and lastly the metric-derived #1 prescription.
  Interventions: Device: Spectacles - Clinically Derived; Device: Spectacles - Metric Technique #1 Derived; Device: Spectacles - Metric Technique #2 Derived
- Metric #1, then Metric #2, then Clinical (Experimental): Each subject will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #1 prescription first, followed by the metric-derived #2 prescription, and lastly the clinically derived prescription.
  Interventions: Device: Spectacles - Clinically Derived; Device: Spectacles - Metric Technique #1 Derived; Device: Spectacles - Metric Technique #2 Derived
- Metric #2, then Metric #1, then Clinical (Experimental): Each subject will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #2 prescription first, followed by the metric-derived #1 prescription, and lastly the clinically derived prescription.
  Interventions: Device: Spectacles - Clinically Derived; Device: Spectacles - Metric Technique #1 Derived; Device: Spectacles - Metric Technique #2 Derived

INTERVENTIONS:
Device: Spectacles - Clinically Derived — Prescription spectacle lenses determined by clinically derived techniques. The specific techniques employed for each subject are left up to the masked examiner and are dependent upon the information needed for refraction determination, as well as ability of the participant to cooperate for testing. Measures may include autorefraction obtained pre or post dilation, retinoscopy obtained pre or post dilation, and subjective refraction obtained pre or post dilation.
  Other Names: Glasses; Prescription Lenses; Spectacles
Device: Spectacles - Metric Technique #1 Derived — Prescription spectacle lenses determined by metric-derived objective technique #1. For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation with the goal of obtaining 3 to 5 high quality captures per eye. Wavefront measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis will then be performed using a computer algorithm to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX). The refractive correction determined from this analysis will be produced in prescription spectacle lenses and dispensed to the patient as the Intervention: Spectacles - Metric Technique #1 Derived.
  Other Names: Glasses; Prescription Lenses; Spectacles
Device: Spectacles - Metric Technique #2 Derived — Prescription spectacle lenses determined by metric-derived objective technique #2. For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation with the goal of obtaining 3 to 5 high quality captures per eye. Wavefront measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis will then be performed using a computer algorithm to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt). The refractive correction determined from this analysis will be produced in prescription spectacle lenses and dispensed to the patient as the Intervention: Spectacles - Metric Technique #2 Derived.
  Other Names: Glasses; Prescription Lenses; Spectacles

SUMMARY:
This study tests the hypothesis that objectively derived spectacle prescriptions based on wavefront aberration measurements of the eyes of individuals with Down syndrome can provide an improvement in visual acuity over that obtained with spectacle prescriptions based on standard clinical prescribing techniques. The objectively derived prescriptions are derived using strategies to optimize retinal image quality as measured by image quality metrics, and thus these prescriptions will be referred to as metric-derived.

DETAILED DESCRIPTION:
Individuals with Down syndrome suffer from significant ocular complications including high levels of lower-order refractive error (sphere and cylinder) and elevated levels of higher-order aberrations. These optical factors likely contribute to the poor acuity observed in this population. Current clinical prescribing practices may under-serve this community, as the cognitive demands of the subjective refraction sequence are difficult for this population and often leave clinicians to prescribe from objective clinical findings that target full correction of sphero-cylindrical refractive error. This prescribing practice can lead to sub-par outcomes given the fact that full lower-order corrections can exacerbate the effects of higher-order aberrations in more aberrated eyes.

For this study, individuals with Down syndrome will be dispensed three pairs of spectacles for 2 months each, in random order: one clinically-derived, and two objectively-derived refractions based upon methods designed to optimize a given metric of retinal image quality which takes into consideration the wavefront aberration measurements of the eye. Both initial and adapted visual acuity in the presence of each correction will be evaluated to determine whether the objectively-derived refractions outperform clinically-derived refractions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome

Exclusion Criteria:

* Nystagmus (Involuntary beating movement of the eyes)
* Visually significant media opacities (e.g. cataracts or corneal scars)
* Strabismic amblyopia (reduced vision in one eye related to a constant eye-turn)
* Anisometropic amblyopia (reduced vision in one eye related to a long-standing uncompensated difference in prescription between the two eyes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Anderson, OD, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Anderson HA, Marsack JD, Benoit JS, Manny RE, Fern KD. Visual Acuity Outcomes in a Randomized Trial of Wavefront Metric-optimized Refractions in Adults with Down Syndrome. Optom Vis Sci. 2022 Jan 1;99(1):58-66. doi: 10.1097/OPX.0000000000001834. PMID 34882603
- [Derived] Anderson HA, Benoit JS, Marsack JD, Manny RE, Ravikumar A, Fern KD, Trast KR. A Randomized Trial of Objective Spectacle Prescriptions for Adults with Down Syndrome: Baseline Data and Methods. Optom Vis Sci. 2021 Jan 1;98(1):88-99. doi: 10.1097/OPX.0000000000001631. PMID 33394936

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical, Then Metric #1, Then Metric #2: Subjects will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the clinically derived prescription first, followed by the metric-derived #1, and lastly the metric-derived #2.
  Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
  Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
  Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
- Clinical, Then Metric #2, Then Metric #1: Subjects will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the clinically derived prescription first, followed by the metric-derived #2, and lastly the metric-derived #1.
  Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
  Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
  Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
- Metric #1, Then Clinical, Then Metric #2: Subjects will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #1 prescription first, followed by the clinically derived, and lastly the metric-derived #2.
  Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
  Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
  Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
- Metric #2, Then Clinical, Then Metric #1: Subjects will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #2 prescription first, followed by the clinically derived, and lastly the metric-derived #1.
  Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
  Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
  Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
- Metric #1, Then Metric #2, Then Clinical: Subjects will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #1 prescription first, followed by the metric-derived #2, and lastly the clinically derived.
  Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
  Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
  Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
- Metric #2, Then Metric #1, Then Clinical: Subjects will receive all three spectacle prescription interventions dispensed in randomized order for 2 months of wear each. Subjects in this arm of the study will receive the metric-derived #2 prescription first, followed by the metric-derived #1, and lastly the clinically derived.
  Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
  Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
  Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
Period: Initial Acuity at Dispense Visit (10min)
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 1 Dispense to 2 Months Wear
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment 2 Dispense to 2 Months Wear
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment 3 Dispense to 2 Months Wear
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed by participant. There was not a unit other than participants assigned to Arms/Groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9) | 30 (13) | 34 (9) | 28 (12) | 24 (4) | 28 (10) | 29 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 3 | 4 | 15
  Male | 2 | 4 | 2 | 4 | 2 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 1 | 2 | 7
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 4 | 3 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 0 | 1 | 4
  White | 3 | 3 | 5 | 3 | 5 | 4 | 23
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 5 | 5 | 30
Adaptive Behavior Standard Score [Median (Full Range); unit: Standard Score] — Participant developmental ability was assessed through the parent/guardian responses on the Vineland 2 Adaptive Assessment. Standard scores <70 indicate low adaptive functioning, scores from 70 to 85 indicate moderately low functioning, and scores from 86 to 115 indicate adequate adaptive function. The total range of possible standard scores on the Vineland is 20 to 160.
  Standard Score | 74 [42 to 99] | 73 [33 to 85] | 59 [22 to 78] | 60 [40 to 79] | 57 [40 to 71] | 59 [54 to 81] | 60 [22 to 99]
Binocular Distance Visual Acuity [Mean (Standard Deviation); unit: logMAR] — Visual Acuity with the participant's presenting correction (or unaided if that had no correction) was obtained with a computerized logMAR style chart with subjects identifying letters from 0.8 logMAR size to progressively smaller sizes in 0.1 logMAR steps (5 letters per line) until a total of 5 mistakes were made. Measures were performed with both eyes open rather than for each eye individually. The potential minimum score on the test (worst vision) was 0.90 logMAR and the potential maximum score (best vision) was -0.20 logMAR.
  logMAR | 0.30 (.10) | 0.48 (0.29) | 0.40 (0.13) | 0.38 (0.15) | 0.46 (0.16) | 0.30 (0.14) | 0.39 (0.17)
Number presenting with spectacles [Count of Participants; unit: Participants] — This is the number of participants who were already wearing prescription spectacles at the time they entered the study.
  Participants | 4 | 4 | 3 | 4 | 2 | 4 | 21
Refractive Error Classification [Number; unit: Number of Eyes] — Refractive error was classified for each eye based on the individual powers of the principal meridians and cylinder magnitude. Myopia was -0.50D or more myopia in both meridians. Hyperopia was a most plus meridian at least +1.00 D with the fellow meridian greater than or equal to 0 D. Mixed astigmatism was one principal meridian with plus power and the other with minus with at least 0.50 D cylinder. Emmetropia was both principal meridians between -0.50 and +1.00 D with less than 0.50 D cylinder.
  Number of Eyes
    Myopia | 5 | 1 | 4 | 1 | 8 | 4 | 23
    Hyperopia | 4 | 6 | 3 | 4 | 1 | 3 | 21
    Mixed Astigmatism | 1 | 3 | 3 | 5 | 0 | 3 | 15
    Emmetropia | 0 | 0 | 0 | 0 | 1 | 0 | 1
Autorefraction Spherical Equivalent OD [Mean (Standard Deviation); unit: Diopters] — Unaided distance autorefraction was performed on the right eye. The spherical equivalent is reported as the spherical power plus 1/2 the cylindrical power.
  Diopters | -1.68 (4.53) | 1.93 (3.07) | -3.73 (7.33) | 0.98 (1.27) | -1.75 (4.37) | -5.23 (4.75) | -1.58 (4.88)
Autorefraction Spherical Equivalent OS [Mean (Standard Deviation); unit: Diopters] — Unaided distance autorefraction was performed on the left eye. The spherical equivalent was calculated as the spherical power plus 1/2 the cylindrical power.
  Diopters | -2.03 (5.91) | 1.95 (2.52) | -2.68 (6.81) | -0.05 (2.43) | -1.58 (4.55) | -3.53 (3.73) | -1.32 (4.59)
Autorefraction Cylinder OD [Mean (Standard Deviation); unit: Diopters] — Unaided distance autorefraction was performed on the right eye. The cylindrical power is reported in minus cylinder form.
  Diopters | -1.45 (0.67) | -3.65 (1.43) | -2.65 (2.91) | -2.25 (1.08) | -1.50 (0.68) | -1.35 (0.68) | -2.14 (1.58)
Autorefraction Cylinder OS [Mean (Standard Deviation); unit: Diopters] — Unaided distance autorefraction was performed on the left eye. The cylindrical power is reported in minus cylinder form.
  Diopters | -1.15 (0.68) | -3.60 (1.32) | -1.55 (1.81) | -2.10 (0.42) | -1.95 (1.45) | -2.05 (0.37) | -2.07 (1.30)

OUTCOME MEASURES:

1. Primary Outcome: Adapted Visual Acuity
Description: Aided LogMAR distance visual acuity obtained with either the British Standard Letters or HOTV - matching for subjects unable to name letters.
Time Frame: two months
Population: Spectacles from the clinical treatment method were not dispensed to one participant in the Metric #1, then Clinical, then Metric #2 group due to failure of the safety criteria required for dispense. This spectacle prescription resulted in visual acuity worse than 7 letters from the participant's presenting acuity to the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
logMAR
  Period 2 Treatment 1 Dispense to 2 Months Wear | 0.256 (0.110) | 0.440 (0.240) | 0.356 (0.149) | 0.284 (0.089) | 0.300 (0.163) | 0.364 (0.048)
  Period 3 Treatment 2 Dispense to 2 Months Wear: number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 5
  Period 3 Treatment 2 Dispense to 2 Months Wear | 0.272 (0.135) | 0.412 (0.215) | 0.370 (0.093) | 0.316 (0.157) | 0.256 (0.344) | 0.316 (0.091)
  Period 4 Treatment 3 Dispense to 2 Months Wear | 0.288 (0.100) | 0.424 (00.238) | 0.320 (0.117) | 0.276 (0.140) | 0.216 (0.119) | 0.372 (0.091)
Statistical Analysis 1: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; It was calculated that 29 participants randomized in a 3x3 within-subject crossover design (repeated measures) achieves at least 89% power to detect an effect size of 0.25. Sample size was determined by a 2-sided f-test (alpha = 0.05) of the overall treatment effect based on a statistical simulation, simulating the repeated measures design. Assumptions included ICC of 0.3; Test type: Other; p = 0.341, Mixed Models Analysis — The threshold for statistical significance was 0.05; f statistic = 1.10
Statistical Analysis 2: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 0.31, 95% CI 2-sided [0.26 to 0.36] — Additional model based estimates for 2-month estimated least square means in binocular visual acuity (logMAR) for PFST
Statistical Analysis 3: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 0.33, 95% CI 2-sided [0.27 to 0.38] — Additional model based estimates for 2-month estimated least square means in binocular visual acuity (logMAR) for VSX
Statistical Analysis 4: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 0.34, 95% CI 2-sided [0.28 to 0.39] — Additional model based estimates for 2-month estimated least square means in binocular visual acuity (logMAR) for Clinical Refraction

2. Secondary Outcome: Initial Visual Acuity
Description: as for outcome 1
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
logMAR
  Treatment 1 Initial Dispense | 0.28 (0.14) | 0.43 (0.25) | 0.34 (0.22) | 0.28 (0.13) | 0.29 (0.35) | 0.33 (0.09)
  Treatment 2 Initial Dispense | 0.25 (0.08) | 0.43 (0.25) | 0.36 (0.18) | 0.30 (0.22) | 0.30 (0.15) | 0.34 (0.07)
  Treatment 3 Initial Dispense | 0.31 (0.40) | 0.44 (0.24) | 0.40 (0.16) | 0.32 (0.18) | 0.28 (0.14) | 0.40 (0.05)
Statistical Analysis 1: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.410, f test — The threshold for statistical significance was 0.05; f statistic = 0.93
Statistical Analysis 2: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 0.35, 95% CI 2-sided [0.28 to 0.41] — Additional model based estimates for initial visit estimated least square means in binocular visual acuity (logMAR) for PFST
Statistical Analysis 3: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 0.33, 95% CI 2-sided [0.26 to 0.39] — Additional model based estimates for initial visit estimated least square means in binocular visual acuity (logMAR) for VSX
Statistical Analysis 4: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 0.34, 95% CI 2-sided [0.28 to 0.41] — Additional model based estimates for initial visit estimated least square means in binocular visual acuity (logMAR) for Clinical Refraction

3. Secondary Outcome: Spectacle Wear Time
Description: Total wear time of each pair of spectacles as measured objectively by a temperature sensor data logger mounted to the spectacle temple.
Time Frame: two months
Population: For Period 3, one participant in group Metric #1, then Clinical, then Metric #2 did not receive the Clinical spectacle treatment because it failed the safety criteria for dispense. The clinical treatment for that participant reduced visual acuity greater than 7 letters from presenting acuity.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Hours
  Period 2 Treatment 1 Dispense to 2 Months Wear | 11.93 (4.95) | 13.15 (3.96) | 10.48 (4.08) | 9.81 (4.32) | 8.40 (4.29) | 11.62 (2.55)
  Period 3 Treatment 2 Dispense to 2 Months Wear: number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 5
  Period 3 Treatment 2 Dispense to 2 Months Wear | 9.50 (5.50) | 12.68 (5.82) | 12.31 (4.74) | 9.67 (4.85) | 9.26 (4.17) | 11.25 (2.96)
  Period 4 Treatment 3 Dispense to 2 Months Wear | 11.61 (6.05) | 13.32 (4.53) | 11.95 (4.18) | 9.47 (5.12) | 9.54 (4.34) | 11.31 (3.06)
Statistical Analysis 1: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.351, f test — The threshold for statistical significance was alpha=0.05; f statistic = 1.09
Statistical Analysis 2: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 11.0, 95% CI 2-sided [9.3 to 12.7] — Additional model based estimates for two-month wear time estimated least square means in spectacle wear-time (Hours) for PFST
Statistical Analysis 3: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 10.9, 95% CI 2-sided [9.2 to 12.6] — Additional model based estimates for two-month wear time estimated least square means in spectacle wear-time (Hours) for VSX
Statistical Analysis 4: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; least square means = 11.2, 95% CI 2-sided [9.5 to 12.9] — Additional model based estimates for two-month wear time estimated least square means in spectacle wear-time (Hours) for Clinical Refraction

4. Secondary Outcome: Spectacle Assessment Survey Question 1
Description: Participants were asked to select a face from a survey with five expressions (large frown, small frown, neutral, small smile, large smile) depicting their response to the question 'Do you like wearing this pair of glasses?' Responses were coded 1 through 5 with 5 = large smile.
Time Frame: two months
Population: A single participant from group 'Metric #1, then Clinical, then Metric #2' was not dispensed the clinical treatment due to the treatment failing one of the safety criteria for dispense.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
score on a scale
  Period 2 Treatment 1 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [2 to 5] | 5 [5 to 5]
  Period 3 Treatment 2 Dispense to 2 Months Wear: number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 5
  Period 3 Treatment 2 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [4 to 5] | 5 [4 to 5] | 4 [4 to 5]
  Period 4 Treatment 3 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 4 [4 to 5]
Statistical Analysis 1: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; It was calculated that a sample size of n=28 yields 82% power to detect a difference of 0.4 in proportion of satisfaction (binary outcome of scores of '4' or '5' versus '1 to 3') in comparing two metrics using a two sided McNemar's test (alpha = 0.025 to account for pairwise testing); Test type: Other; p = 0.562, Mixed Models Analysis; f statistic = 0.58
Statistical Analysis 2: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.967 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 1 for PFST
Statistical Analysis 3: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.933 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 1 for VSX
Statistical Analysis 4: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.897 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 1 for Clinical Refraction

5. Secondary Outcome: Spectacle Assessment Survey Question 2
Description: Participants were asked to select a face from a survey with five expressions (large frown, small frown, neutral, small smile, large smile) depicting their response to the question 'How well do you see with this pair of glasses when looking far away?' Responses were coded 1 through 5 with 5 = large smile.
Time Frame: two months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
score on a scale
  Period 2 Treatment 1 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [4 to 5] | 5 [5 to 5] | 5 [4 to 5] | 5 [5 to 5] | 5 [4 to 5]
  Period 3 Treatment 2 Dispense to 2 Months Wear: number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 5
  Period 3 Treatment 2 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [5 to 5] | 4.5 [4 to 5] | 5 [5 to 5] | 5 [4 to 5] | 4 [4 to 5]
  Period 4 Treatment 3 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [4 to 5] | 5 [5 to 5] | 5 [4 to 5] | 5 [5 to 5] | 5 [5 to 5]
Statistical Analysis 1: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; [analysis description as in outcome 4, analysis 1]; Test type: Other; p > 0.99, Mixed Models Analysis
Statistical Analysis 2: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.967 — Additional estimates of proportion of 2-month satisfactory responses (binary) for 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 2 for PFST
Statistical Analysis 3: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.967 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 2 for VSX
Statistical Analysis 4: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.966 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 2 for Clinical Refraction

6. Secondary Outcome: Spectacle Assessment Survey Question 3
Description: Participants were asked to select a face from a survey with five expressions (large frown, small frown, neutral, small smile, large smile) depicting their response to the question 'How well do you see with this pair of glasses when looking up close?' Responses were coded 1 through 5 with 5 = large smile.
Time Frame: two months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical, Then Metric #1, Then Metric #2 | Clinical, Then Metric #2, Then Metric #1 | Metric #1, Then Clinical, Then Metric #2 | Metric #2, Then Clinical, Then Metric #1 | Metric #1, Then Metric #2, Then Clinical | Metric #2, Then Metric #1, Then Clinical
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
score on a scale
  Period 2 Treatment 1 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [5 to 5] | 5 [4 to 5] | 5 [4 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Period 3 Treatment 2 Dispense to 2 Months Wear: number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 5
  Period 3 Treatment 2 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [5 to 5] | 5 [4.5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Period 4 Treatment 3 Dispense to 2 Months Wear | 5 [5 to 5] | 5 [4 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [4 to 5]
Statistical Analysis 1: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; [analysis description as in outcome 4, analysis 1]; Test type: Other; p > 0.99, Mixed Models Analysis
Statistical Analysis 2: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.967 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 3 for PFST
Statistical Analysis 3: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.967 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 3 for VSX
Statistical Analysis 4: Comparison: Clinical, Then Metric #1, Then Metric #2 vs Clinical, Then Metric #2, Then Metric #1 vs Metric #1, Then Clinical, Then Metric #2 vs Metric #2, Then Clinical, Then Metric #1 vs Metric #1, Then Metric #2, Then Clinical vs Metric #2, Then Metric #1, Then Clinical; Test type: Other; proportion = 0.966 — Additional estimates of proportion of 2-month satisfactory responses (binary) for Spectacle Assessment Survey Item 3 for Clinical Refraction

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of dispense of the first treatment through follow up of the final dispensed treatment (6 months total).
Description: Parents/guardians of participants were contacted by phone one day and one week after each new treatment was dispensed to inquire whether participants were having any difficulty with the glasses. At every visit, participants and their family member were asked if there had been any medical or medication changes since the last visit and if they had any concerns about the spectacles or any new ocular or visual complaints. Reports of glasses needing a fit adjustment were not considered AEs.
Groups:
- Clinical: Spectacles - Clinically Derived: Prescription spectacle lenses determined by clinically derived techniques of a masked examiner and may include autorefraction, retinoscopy, and subjective refraction obtained pre or post dilation.
- Metric #1: Spectacles - Metric Technique #1 Derived: For this method, wavefront error will be measured with the COAS (complete ophthalmic analysis system) wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Visual Strehl ratio in the spatial domain (VSX).
- Metric #2: Spectacles - Metric Technique #2 Derived: For this method, wavefront error will be measured with the COAS wavefront aberrometer post-dilation (3 - 5 captures per eye). Measures will be re-sized to the patient's habitual pupil diameter and averaged. Post-measurement analysis is performed to identify the refractive correction predicted to produce the best image quality, as measured by maximization of the image quality metric Pupil Fraction tessellated (PFSt).
Arm/Group | Clinical | Metric #1 | Metric #2
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 7/29 | 5/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical (N=29) | Metric #1 (N=30) | Metric #2 (N=30)
Vision complaint related to comparison with earlier randomized treatment or habitual spectacles (Eye disorders) | 7 (7) | 1 (1) | 2 (2) — Patients reporting blur at a particular viewing distance, not liking glasses as well as previous ones, or changing glasses wear behavior.
Upper Respiratory Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 2 (3) — Reports of cough or runny nose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03367793/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT03367793/SAP_001.pdf